CLINICAL TRIAL: NCT04187560
Title: A Randomized, Double-blinded, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LB-102 Administered Orally to Healthy Subjects
Brief Title: Safety and Tolerability of Single and Multiple Doses of LB-102 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LB Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: LB-102-001
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A Cohort 1 (Active Comparator): LB-102 50 mg (n=6) or Matching Placebo (n=2) x 1 day
  Interventions: Drug: LB-102
- Part A Cohort 2 (Active Comparator): LB-102 15 mg (n=6) or Matching Placebo (n=2) x 1 day
  Interventions: Drug: LB-102
- Part A Cohort 3 (Active Comparator): LB-102 100 mg (n=6) or Matching Placebo (n=2) x 1 day
  Interventions: Drug: LB-102
- Part A Cohort 4 (Active Comparator): LB-102 200 mg (n=6) or Matching Placebo (n=2) x 1 day
  Interventions: Drug: LB-102
- Part A Cohort 5 (Active Comparator): LB-102 150 mg (n=6) or Matching Placebo (n-2) x 1 day
  Interventions: Drug: LB-102
- Part B Cohort 6 (Active Comparator): LB-102 50 mg (n=6) or Matching Placebo (n=2) BID x 7 days (QD on Day 7)
  Interventions: Drug: LB-102
- Part B Cohort 7 (Active Comparator): LB-102 100 mg (n=6) or Matching Placebo (n=2) BID x 7 days (QD on Day 7)
  Interventions: Drug: LB-102
- Part B Cohort 8 (Active Comparator): LB-102 75 mg (n=6) or Matching Placebo (n=2) BID x 7 days (QD on Day 7)
  Interventions: Drug: LB-102

INTERVENTIONS:
Drug: LB-102 — (N-Methyl amisulpride)
  Other Names: Active Drug

SUMMARY:
A Single Ascending Dose (SAD; Part A) and Multiple Ascending Dose (MAD; Part B) Phase 1 Study of LB-102 N-Methyl amisulpride) in healthy volunteers. The primary objective is to evaluate the safety and the tolerability of a single oral dose (SAD) and multiple oral doses (MAD) of LB-102 as compared to placebo. The secondary objectives are to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of LB-102.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled study designed to evaluate the safety, tolerability, and pharmacokinetics of LB-102 in healthy subjects. The study will consist of two parts: Part A - Single Ascending Dose and Part B - Multiple Ascending Doses. There will be 5 cohorts in Part A and 3 Cohorts in Part B of this study. Each cohort consists of 8 subjects, with 6 subjects assigned to LB-102 and 2 subjects assigned to placebo.

In Parts A and B, eligible subjects will be randomized on Day 1 (pre-dose) to placebo (n=2) or LB-102 (n=6). Eligible subjects will receive 1 dose on Day 1 (Part A) or 13 doses on Days 1-7 (Part B) of placebo or LB-102.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study only if they meet all of the following criteria:

1. Competent to provide informed consent.
2. Voluntarily provide informed consent.
3. Healthy adult male and female subjects between 18 to 55 years of age inclusive at the screening visit.
4. Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m2 at screening visit.
5. Subjects must be in good general health as determined by medical history and physical examination with no clinically significant medical findings and no history of significant medical disease (e.g. cardiovascular, pulmonary, renal, etc.) or acute condition with the past 30 days.
6. Have normal clinical laboratory test results and ECG, which are not considered to be clinically significant by the investigator.
7. Female subjects of child-bearing potential must agree to use two methods of an acceptable method of birth control (e.g., condom and spermicide, intrauterine device (IUD), oral contraception which has been stable for 30 days) and at least 90 days after stopping the investigational product. Female subjects using oral contraception whose partner consistently uses condoms or who is vasectomized is also acceptable.
8. Male subjects must be surgically sterile or practicing at least one method of contraception, from initial study drug administration through 90 days after administration of the last dose of study drug:
9. Male subjects must agree to abstain from sperm donation through 90 days after administration of the last dose of investigational drug.

Exclusion Criteria:

Subjects will be excluded from the study for any of the following reasons:

1. Are pregnant or lactating.
2. Have a history or presence of significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorders which, in the opinion of the investigator, increases the risk of the study drug or may confound the interpretation of study measures.
3. Clinically significant abnormal findings on physical examination, vital signs, or ECG.
4. History or presence of psychiatric or neurological disease or condition.
5. History of seizures.
6. Subject with any history or current evidence of suicidal behavior.
7. Unwilling to complete any planned study assessments, including the Columbia-Suicide Severity Rating Scale (CSSRS).
8. Recent history of alcohol or drug abuse (within the last two years).
9. Any use of tobacco or tobacco-containing products (cigarettes, pipes, etc.) within one month prior to screening.
10. Have a history of blood donation in excess of 500 mL of blood within 30 days prior to Screening.
11. Have received treatment with an investigational drug or device within 30 days prior to Screening.
12. Use of any prescription or over the counter medication, herbal medications, vitamins, or supplements within 14 days prior to study drug administration.
13. Have a positive test for human immunodeficiency virus (HIV) antibodies 1 and 2, Hepatitis B surface antigen or Hepatitis C antibody.
14. Any subject who is known to be allergic to the study drug or any components of the study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who experience at least one treatment-emergent adverse event (TEAE) | Day 8 (Part A) or Day 15 (Part B)
  A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A TEAE may also be a pre-treatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug, which increases in intensity after the start of dosing.

SECONDARY OUTCOMES:
Tmax: Time to Reach the Maximum Plasma Concentration | Days 1, 2 and 3 (Part A) Days 1 through 9 (Part B)
  Time to reach the maximum observed plasma concentration for LB-102 and LB-102 metabolite amisulpride after a single dose (Day 1) and multiple dosing (Day 7).
Cmax: Maximum Observed Plasma Concentration | Days 1, 2 and 3 (Part A) Days 1 through 9 (Part B)
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Cmax will be measured for LB-102 and LB-102 metabolite amisulpride after a single dose (Day 1) and multiple dosing (Day 7).
AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration | Days 1, 2 and 3 (Part A) Days 1 through 9 (Part B)
  AUC(0-tlqc) is a measure of total plasma exposure to a drug from time 0 to time of the Last Quantifiable Concentration and will be measured for LB-102 and LB-102 metabolite amisulpride after a single dose (Day 1) and multiple dosing (Day 7)
AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose | Days 1, 2 and 3 (Part A) Days 1 through 9 (Part B)
  AUC(0-24) is a measure of total plasma exposure to the drug from Time 0 to 24 hours post-dose for LB-102 and LB-102 metabolite amisulpride after a single dose (Day 1) and multiple dosing (Day 14).

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Biernat, MD, Principal Investigator — Medpace, Inc.
Locations (1):
- Medpace Clinical Pharmacology LLC, Cincinnati, Ohio, United States

REFERENCES:
- See also: Corporate Website — http://www.LBPharma.us
- Available data/document: Clinical Study Report — http://lbpharma.us/wp-content/uploads/2020/12/lb-102-001-clinical-study-report-final.pdf